CLINICAL TRIAL: NCT01280825
Title: The 1200 Patients Project: Studying the Implementation of Clinical Pharmacogenomic Testing
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 10-487-A
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Patients Undergoing Routine Health Care; Heart Diseases; Inflammatory Bowel Diseases; Autoimmune Disease; Inflammatory Disease; Blood Coagulation Disorders; Hepatitis C; Non-Metastatic Neoplasm
MeSH Terms: conditions — Heart Diseases; Inflammatory Bowel Diseases; Autoimmune Diseases; Blood Coagulation Disorders; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult Patients: Adults receiving health care at the University of Chicago Medical Center.

SUMMARY:
The purpose of this study is to collect DNA samples from patients undergoing routine care at the University of Chicago. These samples will be tested for differences in genes that may suggest greater risk of side effects or chance of increased benefit from certain medications. The results will be made available to the patient's treating physician and the researchers will track whether or not this information is used in routine health care.

ELIGIBILITY:
Inclusion Criteria:

* Receiving ongoing, out-patient care at the University of Chicago Medical Center under the routine care of a physician participating in this trial
* Life expectancy of at least 3 years
* Must be 18 years or older
* Must be taking at least 1 (but not more than 6) prescription medications at the time of enrollment OR be 65 years or older OR be reasonably expected to require the use of a prescription medication within the next 5 years
* Patients with certain diseases, or likely to receive or be receiving certain drugs, will be targeted particularly for enrollment in order to enrich the study for patients likely to have pharmacogenetically relevant interactions, including, but not limited to:

  * Patients requiring specialized cardiology care
  * Patients with inflammatory bowel diseases
  * Patients with systemic autoimmune or inflammatory diseases
  * Patients requiring long-term oral anticoagulation
  * Patients with hepatitis C
  * Patients with non-metastatic cancer

Exclusion Criteria:

* Patients with acute or chronic disease which could be reasonably expected to result in the patient's death within the next 3 years.
* Patients who have undergone, or are being actively considered for, liver or kidney transplantation.
* Inability to understand and give informed consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults receiving ongoing routine medical care and regularly using at least 1 (but no more than 6) prescription medications at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2011-01-14 (Actual); Primary Completion 2027-11-14 (Estimated); Study Completion 2027-12-14 (Estimated)

PRIMARY OUTCOMES:
Feasibility of incorporating pharmacogenomic testing into routine medical care | 5 years

SECONDARY OUTCOMES:
Find out whether availability of pharmacogenomic information impacts drug decision making in the health care setting | 5 years

OTHER OUTCOMES:
To determine whether access to pharmacogenomic information improves satisfaction with care. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter H O'Donnell, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States